CLINICAL TRIAL: NCT00474500
Title: Effect of Coca-Cola on Iron Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: University of East Anglia (Other); The Coca-Cola Company (Industry)
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IFR13/2006
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Iron Deficiency
Keywords: Iron absorption; Coca-Cola
MeSH Terms: conditions — Iron Deficiencies | interventions — Cocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Coca, Cola, Diet Coke

SUMMARY:
The aim of this project is to measure the effect of Coca-Cola and Diet Coke, relative to mineral water, on non-haem iron absorption. The results from this study will quantify any enhancing effect of Coca-Cola or Diet Coke on non-haem iron absorption and will be of use to the Coca-Cola Company and the scientific and nutrition community in evaluating the nutritional value of these products.

DETAILED DESCRIPTION:
Previous studies have suggested that Coca-Cola may enhance absorption of non-haem iron. A randomized cross-over trial will be undertaken to compare the absorption of iron added to a pizza meal consumed with either Coca-Cola, Diet Coke or mineral water. Pizza containing added iron, labelled with an iron stable isotope (Fe-58), will be consumed for lunch on two consecutive days with either a Coca-Cola, Diet Coke or mineral water drink. Iron absorption from the pizza will be determined using the erythrocyte incorporation technique.

A baseline blood sample will be taken prior to consuming the first test meal (pizza + drink 1) and after approximately 15 days, a second fasting blood sample will be taken prior to consumption of a second set of test meals (pizza + drink 2). Iron isotope enrichment of the blood sample will be used as a baseline for the second set of test meals and to calculate absorption from the first set of test meals. A third blood sample will be taken after approximately 30 days and the iron isotope enrichment will be used as a baseline for the third set of test meals (pizza + drink 3) and to determine absorption from the second set of test meals. At about 45 days a final blood sample will be taken to determine absorption from the third set of test meals. Iron absorption will be calculated from the isotopic enrichment in blood, assuming that 80% of absorbed iron is incorporated into red blood cells. Absorption of iron consumed with Coca-Cola and Diet Coke will be compared with iron absorption when consumed with mineral water. The order in which the volunteers will be given the drinks will be randomised.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age > 18 and < 65

Exclusion Criteria:

* Men
* Age < 18 or > 65
* BMI <18.5 or > 35
* Serum ferritin value of <12 or >50µg/L (±10% to allow for day to day and analytical variation)
* Volunteers will be excluded if they are found to have depressed or elevated blood pressure measurements (<90/50 or <95/55 if symptomatic or >160/100)
* Diagnosed with a long-term illness requiring active treatment, e.g. diabetes, cancer, cardiovascular disease.
* Gastrointestinal disease (excluding hiatus hernia unless symptomatic or study intervention/procedure is contraindicated)
* Regular prescribed medication that may interfere with iron metabolism
* Regular use of antacids and laxatives (at least once a week)
* Women who are pregnant or less than 12 months since giving birth
* Women breast feeding
* Vitamin supplements with or without minerals if taken more than once a week, and unwillingness to discontinue occasional use for the duration of study
* Unwillingness to discontinue use of herbal supplements for the duration of study
* Use of antibiotics within four weeks prior to study start
* Parallel participation in another study which involves dietary interventions or sampling of blood that may increase the volume taken above 500ml in a 4-month period
* Asthma requiring treatment within the last two years
* Results of clinical screening which indicate, or are judged by the HNU Medical Advisor to be indicative of a health problem which could compromise the well-being of the volunteer if they participated or which would affect the study data.
* Allergy to any of the ingredients in the test meals

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Non-haem iron absorption | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Fairweather-Tait, Principal Investigator — University of East Anglia
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Collings R, Fairweather-Tait SJ, Dainty JR, Roe MA. Low-pH cola beverages do not affect women's iron absorption from a vegetarian meal. J Nutr. 2011 May;141(5):805-8. doi: 10.3945/jn.110.136507. Epub 2011 Mar 9. PMID 21389184